CLINICAL TRIAL: NCT06908772
Title: A Multicenter Phase II/III Clinical Study on the Efficacy and Safety of Glumetinib Combined With Osimertinib as First-Line Treatment in Non-Small Cell Lung Cancer Patients With Classical EGFR Mutations Accompanied by MET Amplification or Overexpression
Brief Title: Glumetinib Combined With Osimertinib Treatment for Non-Small Cell Lung Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYH2065-003
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Recurrent or Metastatic NSCLC Patients With Classical EGFR Mutations Accompanied by MET Amplification or Overexpression
MeSH Terms: conditions — Recurrence | interventions — glumetinib; osimertinib

STUDY DESIGN:
Intervention Model Description: Randomized, positive-controlled Phase Ⅱ/Ⅲ
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Glumetinib（200 mg） + Osimertinib (Experimental): Group 1: Glumetinib 200 mg oral QD + Osimertinib 80 mg oral QD.
  Interventions: Drug: Glumetinib Tablets; Drug: Osimertinib Mesylate Tablets
- Glumetinib（300mg） + Osimertinib (Experimental): Group 2: Glumetinib 300 mg oral QD + Osimertinib 80 mg oral QD;
  Interventions: Drug: Glumetinib Tablets; Drug: Osimertinib Mesylate Tablets
- Osimertinib (Experimental): Group 3: Osimertinib 80 mg oral QD.
  Interventions: Drug: Osimertinib Mesylate Tablets; Drug: Glumetinib Tablets Placebo

INTERVENTIONS:
Drug: Glumetinib Tablets — An ATP competitive, highly selective MET receptor tyrosine kinase inhibitor
  Arms: Glumetinib（200 mg） + Osimertinib; Glumetinib（300mg） + Osimertinib
Drug: Osimertinib Mesylate Tablets — 3rd EGFR-TKI
Drug: Glumetinib Tablets Placebo — Placebo
  Arms: Osimertinib

SUMMARY:
To evaluate the efficacy and safety of glumetinib combined with osimertinib as the first-line treatment for locally advanced or metastatic NSCLC.

DETAILED DESCRIPTION:
In the Phase II stage, eligible subjects who have passed screening will be randomly assigned in a 1:1:1 ratio into the Group 1, Group 2, and Group 3 to receive study treatment:

In the Phase III stage, eligible subjects who have passed screening will be randomly assigned in a 1:1 ratio into the test group and the control group to receive the study treatments, and the RP3D obtained from Phase II will be used as the dose of glumetinib for the test group.

Randomization stratification factors include: c-MET status (≥2+, ≥75% and 3+, <50% vs 3+, ≥50% or FISH positive), and EGFR-sensitive mutation type (19Del vs L858R).

In both the Phase II and Phase III stages, each treatment cycle is every 3 weeks, with continuous treatment until progressive disease (PD) confirmed by the investigator, intolerable toxicity, withdrawal of informed consent by the subject, loss to follow-up, death, or other criteria for terminating treatment as specified in the protocol, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to understand and voluntarily sign the written informed consent form (ICF); 2. Male or female subjects aged 18 to 75 years (inclusive). 3. Patients with NSCLC who have unresectable locally advanced or metastatic disease; 4. At least one measurable lesion, as defined by RECIST 1.1 criteria; 5. ECOG performance status of 0 or 1; 6. Expected survival ≥ 3 months; 7. Adequate function of major organs and bone marrow; 8. Women or man of childbearing potential must use highly effective contraception.

Exclusion Criteria:

1. Prior treatment with an EGFR inhibitor or MET inhibitor;
2. Patients with metastases to meninges; with spinal cord compression; symptomatic and unstable brain metastasis;
3. Patients who have taken strong inducers or inhibitors of CYP3A4 within 2 weeks prior to the first dose of the study drug, or who cannot discontinue the use of strong CYP3A4 inducers and inhibitors during the study;
4. Patients with a history of autoimmune diseases, a history of immunodeficiency, including positive for HIV, or other acquired or congenital immunodeficiency diseases, or a history of organ transplant;
5. Presence of active infection (e.g., subjects are receiving anti-infection therapy);
6. Severe or uncontrolled cardiovascular disorder requiring treatment;
7. Refractory nausea, vomiting, chronic gastrointestinal disease, inability to swallow drugs orally;
8. Women who are pregnant or breastfeeding;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Phase 2：ORR as assessed by IRC | Up to approximately 30 months after the first participant is enrolled

SECONDARY OUTCOMES:
Phase 2：ORR as assessed by investigator | Up to approximately 30 months after the first participant is enrolled
phase 2：PFS as assessed by IRC and investigator | Up to approximately 30 months after the first participant is enrolled
Phase 3：PFS as assessed by invetigator | Up to approximately 30 months after the first participant is enrolled
Phase 3：ORR as assessed by IRC and investigator | Up to approximately 30 months after the first participant is enrolled
phase 2/3：OS | Up to approximately 30 months after the first participant is enrolled
phase 2/3：DCR as assessed by IRC and investigator | Up to approximately 30 months after the first participant is enrolled
phase 2/3：DoR as assessed by IRC and investigator | Up to approximately 30 months after the first participant is enrolled
phase 2/3：TTR as assessed by IRC and investigator | Up to approximately 30 months after the first participant is enrolled
phase 2/3：Frequency and severity of AEs (NCI CTCAE 5.0) | Up to approximately 30 months after the first participant is enrolled
phase 2/3：PK parameters: The plasma concentration of glumetinib | Up to approximately 30 months after the first participant is enrolled
phase 2/3：Biomarkers: c-MET expression and amplification levels, tumor-related gene mutations | Up to approximately 30 months after the first participant is enrolled

IPD SHARING:
Plan to Share IPD: No